CLINICAL TRIAL: NCT02470104
Title: A Randomized Study of Enteral Donor Human Milk in Young Children Receiving Bone Marrow Transplantation
Brief Title: Donor Human Milk in Young Children Receiving Bone Marrow Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Prolacta Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-4127
Record Dates: First submitted 2015-04-01; First posted 2015-06-12 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Bone Marrow Transplant - Autologous or Allogeneic
Keywords: children; bone marrow transplant; autologous; allogeneic; breastmilk; hematopoietic stem cell transplantation (HSCT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral Donor Breastmilk (Experimental): * Donor milk will be pasteurized prior to use.
  * Given orally or by nasogastric (NG) or nasojejunal (NJ) tube.
  * Feeding will be supervised and will be advanced as quickly as tolerated with a goal of providing 40-50% of nutritional needs from the donor milk.
  * It is recognized that the volume of enteral feeds will need to be adjusted per patient tolerance.
  Interventions: Dietary Supplement: Breastmilk
- Control (No Intervention): • Children randomized to the control arm will receive standard enteral or parenteral nutrition per standard clinical practice, supervised by a registered dietician.

INTERVENTIONS:
Dietary Supplement: Breastmilk — * A registered dietician will supervise milk provision.
  * If a nursing mother enrolls on the study, maternal and not donor milk will be given in the maximum volume possible with Prolacta supplementation if clinically indicated and recommended by the registered dietician.
  Arms: Enteral Donor Breastmilk

SUMMARY:
The investigators hypothesize that children receiving human milk will maintain a greater diversity of helpful bacteria in their gut and have lower levels of inflammatory proteins in the blood compared with children not receiving human milk.

DETAILED DESCRIPTION:
The investigators hypothesize that the gut microbiota during bone marrow transplant could be influenced by administration of enteral donor breast milk. This study will attempt to address this hypothesis, by feeding donor breast milk to young children undergoing transplant, and serially comparing the gut microbiota in children receiving human milk, with those receiving conventional feeding.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 5 years old receiving transplant (autologous or allogeneic)
* Parents must give informed consent

Exclusion Criteria:

* Failure to meet inclusion criteria

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05-25 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Percentage of lactobacillales | 21 days after transplant
  Bar chart to indicate percentage of lactobacillales in stool samples.

SECONDARY OUTCOMES:
Pro-inflammatory cytokine level | weekly during study course; up to approximately one year
  Mean fold increase above baseline for the cytokine will be calculated and compared to control. Value will be tested for statistical significance using the Wilcoxon Rank Sum test.
Incidence of bacteremia | though day 14 post transplant
  Frequency of bacterial sepsis to be compared against controls.
Incidence of graft versus host disease (GVHD) | through study course; approximately one year
  Frequency of GVHD will be compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MB.BS, PhD, MRCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States